CLINICAL TRIAL: NCT04520594
Title: OptiMized REsistaNt Starch in Inflammatory Bowel Disease: The MEND Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, David Mack, Director, CHEO IBD Centre, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 20/16E
Record Dates: First submitted 2020-07-31; First posted 2020-08-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease; Ulcerative Colitis; Inflammatory Bowel Diseases
Keywords: Resistant Starch; Microbiome
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Resistant Starch

STUDY DESIGN:
Intervention Model Description: A single center, randomized, placebo-controlled, double-blinded, parallel, pilot clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unblinding will occur only if necessary to ensure study participants safety, interim analysis at 5 ± 1 months, or eligibility for our associated open label trail (OARS trial). Only Dr. Mack (Co-PI) can request to break the blind for safety reasons or eligibility for the OARS Trial; only Dr. Stintzi (Co-PI) will request to break the blind for interim analysis. Once the blind is broken, the patient will be discontinued from study product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistant Starch (Active Comparator): Once daily oral consumption of 7.5g/m2 of an individually optimized resistant starch for approximately 6 months
  Interventions: Other: Resistant Starch
- Placebo (Placebo Comparator): Once daily oral consumption of a food-grade cornstarch that is readily digestible for approximately 6 months
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Resistant Starch — 7.5 g resistant starch/m2 oral consumption
  Arms: Resistant Starch
Other: Placebo — Placebo oral consumption of food-grade cornstarch
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine if a plant-based resistant starch that is optimized for the individual will target the underlying cause of inflammatory bowel disease and restore a "healthier" gut microbiome in pediatric participants with inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent, or if appropriate, have an acceptable representative capable of giving consent on the participant's behalf.
* Enrolled in the main parent study.
* Existing Crohn's disease or ulcerative colitis diagnosis.
* In clinical remission or with mild disease (wPCDAI of 0-39.5 for CD; PUCAI of 0-30 for UC) with no changes in standard of care treatment for the previous month and without anticipated changes for the next month.
* Ability and willingness to comply with study procedures (e.g. stool collections) for the entire length of the study.
* Willing to provide consent/assent for the collection of stool samples.

Exclusion Criteria:

* Allergy to resistant starch or excipients.
* Co-existing diagnosis with diabetes mellitus.
* Treatment with another investigational drug or intervention throughout the study.
* Current drug or alcohol dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of an individual or legal guardian to give written informed consent.
* Concomitant chronic disease requiring medications.
* Requirement for antibiotic therapy >2 weeks duration.
* Participant's microbiota does not respond to any of the resistant starch from the assembled panel as measured through the RapidAIM evaluation following the initial stool sample collection.
* Patients with previous intestinal surgery.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Increased potential of butyrate production following the use of individualized resistant starch, as assessed by meta-omics analysis. | 6 ± 1 months
Sustained potential for butyrate production following 6 months use of individualized resistant starch post randomization as assessed by meta-omics analysis. | 12 ± 2 months
Change in microbiome composition of cases towards the microbiome of controls as assessed by meta-omics analysis. | 6 ± 1 months and 12 ± 2 months

SECONDARY OUTCOMES:
Changes in patient reported disability outcomes as measured by the IBD Disability Index Questionnaire. | Enrollment, 3 ± 1 months, 6 ± 1 months , 9 ± 1 months and 12 ± 2 months
  The IBD disability index consists of 28 questions and a higher overall score is indicative of greater disability.
Changes in patient, parent/caregiver reported quality of life outcomes as measured by the IMPACT III Questionnaires. | Enrollment, 3 ± 1 months, 6 ± 1 months , 9 ± 1 months and 12 ± 2 months
  The IMPACT III questionnaire (a health related quality of life questionnaire) consists of 35 questions and ranges in score from 0 to 231. A higher score represents a higher quality of life. The IMPACT III-P Questionnaire is to be completed by the caregiver/guardian with a higher score also representing a higher quality of life.
Changes in intestinal mucosal inflammation by measuring fecal calprotectin through stool samples. | Enrollment, 3 ± 1 months, 6 ± 1 months, 9 ± 1 months, and 12 ± 2 months
Change in clinical disease activity as measured by the wPCDAI for Crohn's Disease. | Enrollment, 3 ± 1 months, 6 ± 1 months , 9 ± 1 months and 12 ± 2 months
  Weighted Pediatric Crohn's Disease Activity Index (wPCDAI) ranges from 0 to 125 points (<12.5 = remission, 12.5 to 40.0 = mild, >40.0 = moderate, >57.5 = severe).
Change in clinical disease activity as measured by the PUCAI for Ulcerative Colitis. | Enrollment, 3 ± 1 months, 6 ± 1 months , 9 ± 1 months and 12 ± 2 months
  The Pediatric Ulcerative Colitis Activity Index (PUCAI) ranges from 0 to 85 points (<10 = remission, 10 to 34 = mild, 35 to 64= moderate, >65 = severe).
Change in clinical disease activity as measured by the Partial Mayo Score for Ulcerative Colitis. | Enrollment, 3 ± 1 months, 6 ± 1 months , 9 ± 1 months and 12 ± 2 months
  The Partial Mayo Score ranges from 0 to 9 points (0 to 1 = remission, 2 to 4 = mild, 5 to 6 = moderate, 7 to 9 = severe).
Change in clinical disease activity as measured by the PGA for both Crohn's Disease and Ulcerative Colitis. | Enrollment, 3 ± 1 months, 6 ± 1 months , 9 ± 1 months and 12 ± 2 months
  The Physician Global Assessment (PGA) ranges from 0 to 3 points (0 = normal, 1 = mild, 2 = moderate, 3 = severe).

CONTACTS AND LOCATIONS:
Overall Officials: David Mack, MD, FRCPC, Principal Investigator — Children's Hospital of Eastern Ontario; Alain Stintzi, PhD, Principal Investigator — University of Ottawa
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada